CLINICAL TRIAL: NCT05985993
Title: Precise Intervention Technology and Application of Low Intensity Transcranial Ultrasound Stimulation (TUS) on Negative Symptoms of Schizophrenia
Brief Title: Precise Intervention Technology and Application of Low Intensity TUS on Negative Symptoms of Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022JC009
Record Dates: First submitted 2023-07-17; First posted 2023-08-14 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-11

CONDITIONS: Negative Symptoms of Schizophrenia
Keywords: Schizophrenia; Negative Symptoms; Transcranial Ultrasound Stimulation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- single-target group (left DLPFC) (Active Comparator): 27 eligible patients will be treated with active TUS for 4 weeks on the left DLPFC
  Interventions: Device: low-intensity transcranial ultrasound stimulation (TUS)
- both-target group (both left DLPFC and right STG) (Active Comparator): 27 eligible patients will be treated with active TUS for 4 weeks on the both left DLPFC and right STG
  Interventions: Device: low-intensity transcranial ultrasound stimulation (TUS)
- sham group (Sham Comparator): 27 eligible patients will be treated with sham TUS for 4 weeks on the left DLPFC and right STG, respectively.
  Interventions: Device: low-intensity transcranial ultrasound stimulation (TUS)

INTERVENTIONS:
Device: low-intensity transcranial ultrasound stimulation (TUS) — The rTUS was administered using an immersion-type focused ultrasound transducer (V391-SU, Olympus NDT, Waltham, USA). Low-intensity transcranial ultrasound stimulation on the target. Duration:20 days (workdays for four consecutive weeks).

SUMMARY:
Based on the current background and our previous studies, TUS has been proved that rTUS intervention could induce long-term potentiation like (LTP-like) plasticity and neuromodulate the brain cortex in schizophrenia patients. rTUS over the left dorsolateral prefrontal cortex (DLPFC) can alleviate the negative symptoms in schizophrenia. In this double-blind, randomized, sham-controlled study, the efficacy of different treatment options and mechanisms of low-intensity rTUS on negative symptoms will be investigated.

DETAILED DESCRIPTION:
Negative symptoms is a core symptom of schizophrenia related to poor functional outcome which remains largely treatment refractory. Prior studies indicated that abnormalities in the prefrontal-temporal circuit and glutamate/GABA imbalances may be the root causes of negative symptoms. Transcranial ultrasound stimulation (TUS), an emerging non-invasive neuromodulation technique, can modulate neuroplasticity in the prefrontal and temporal cortex. In this double-blind, randomized, sham-controlled study, the efficacy of different treatment options and mechanisms of low-intensity rTUS on negative symptoms will be investigated. Schizophrenia inpatients with predominant negative symptoms will be recruited and randomly allocated into single-target group (left DLPFC), both-target group (both left DLPFC and right STG) or sham group in ratio of 1:1:1. This study aims to determine the efficacy of TUS and to reveal its underlying neural mechanism. MEPs, TEPs ,multi-modal MRI and rs-EEG will be detected. Neuropsychological assessments will also be conducted to develop the optimized treatment strategy. The study points to a novel and promising therapeutic neuromodulation approach that may improve the functional outcome of schizophrenia, which has been the main cause of mental disability.

ELIGIBILITY:
Inclusion Criteria:

* Meet the DSM-5 diagnostic criteria for schizophrenia or schizoaffective disorder;
* Age18-50, right-handed, Han nationality;
* Score of at least 1 item from N1 to N7 in PANSS is ≥4 (moderate or above);
* Be in a stable condition, received second-generation antipsychotics for at least 4 weeks or more;
* Written informed consent;

Exclusion Criteria:

* Current or past neurological illness, severe physical diseases, substance abuse or alcohol dependence, mental retardation, pregnant or lactation;
* Uncooperative or risky patients with high excitement, stupor, disorder of words and deeds, negative suicide, etc.;
* History of MECT or other physical therapy within 6 months;
* History of epilepsy, or epileptic waves on the baseline EEG;
* Ruled out share antiepileptic drugs, carbamazepine, valproic acid salt) or larger doses of benzodiazepines drugs (> 10 mg/day, diazepam clonazepam 2 mg/day, 1 mg/day, alprazolam lorazepam 2 mg/day, midazolam 10 mg/day, 20 mg/day, Mr Shah diazepam triazolam 0.5 mg/day), avoid the use of chlorine drug, (in principle, to avoid the use of antiepileptic drugs and clonazepam;Other antipsychotic drugs, if necessary, remain unchanged during the course of treatment;
* Contraindications to TUS and MRI are present.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Brief Negative Symptom Scale (BNSS) | baseline, 4 weeks and 8 weeks
  Change from baseline in the Brief Negative Symptom Scale (BNSS) at 4 weeks and 8 weeks. The minimum to maximum value is 0-78. Lower scores mean a better outcome.
Change from baseline in the Scale for Assessment of Negative Symptoms(SANS) | baseline, 4 weeks and 8 weeks
  Change from baseline in the Scale for Assessment of Negative Symptoms(SANS) at 4 weeks and 8 weeks. The minimum to maximum value is 0-120. Lower scores mean a better outcome.
Change from baseline in Positive and Negative Syndrome Scale(PANSS) | baseline, 4 weeks and 8 weeks
  Change from baseline in Positive and Negative Syndrome Scale(PANSS) at 4 weeks and 8 weeks. The minimum to maximum value is 30-210. Lower scores mean a better outcome.

SECONDARY OUTCOMES:
Change of cognitive Function | baseline, 4 weeks and 8 weeks
  Change from baseline in MATRICS MCCB
Change of Multi-modal Brain Neuroimaging in structure | baseline and 4 weeks
  Brain structure data will be acquired.
Change of Multi-modal Brain Neuroimaging in resting- state fMRI | baseline and 4 weeks
  Resting-state fMRI data will be acquired.
Change of Multi-modal Brain Neuroimaging in 1H-MRS | baseline and 4 weeks
  1H-MRS data will be acquired.
Change of EEG microstates | baseline and 4 weeks
  EEG microstates propose that resting-state neural activity is characterized by several globally functional states with specific spatial distributions at sub-second temporal scales. In this study, resting-state 64-channel EEG data were collected from participants before and after rTUS treatment (at baseline and 4 weeks). The aim was to investigate the effects of rTUS on seven types of EEG microstates in individuals with schizophrenia, as well as the association between changes in temporal parameters and psychiatric symptoms before and after treatment. This study seeks to evaluate the overall brain function and temporal dynamics in schizophrenia, as well as the impact of rTUS intervention on the temporal parameters of different microstates.
Change of TEPs | baseline, Day1, and 4weeks
  TMS-evoked potentials (TEPs) from two target regions (the left DLPFC and the right STG) were measured in participants at baseline, after a single TUS intervention, and at 4 weeks. The study aimed to clarify the effects of rTUS treatment on the components of TEPs in individuals with schizophrenia, as well as the association between changes in TEP components and psychiatric symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No